CLINICAL TRIAL: NCT06750432
Title: A Phase 1b, Double-Blind, Placebo-Controlled, Multiple Ascending Dose Study of the Safety, Tolerability, Pharmacokinetics, Pharmacodynamics, and Preliminary Efficacy of PMN310 in Patients With Early Alzheimer's Disease
Brief Title: PMN310 in Patients With Early Alzheimer's Disease (PRECISE-AD)
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: ProMis Neurosciences, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: PMN310-102
Record Dates: First submitted 2024-12-16; First posted 2024-12-27 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Alzheimer Disease, Early Onset
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Intervention Model Description: There will be 3 sequential escalating dose cohort groups. Dose groups are 350 mg, 700 mg, and 1400 mg administered as a single 60-minute infusion.
Who Masked: Participant, Investigator
Masking Description: Double bind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Cohort 1 PMN310 350 mg or placebo (Experimental): PMN310 350 mg or placebo administered as a 60-minute infusion.
  Interventions: Drug: PMN310; Drug: Placebo
- Cohort 2 PMN310 700 mg or placebo (Experimental): PMN310 700 mg or placebo administered as a 60-minute infusion.
  Interventions: Drug: PMN310; Drug: Placebo
- Cohort 3 PMN310 1400 mg or placebo (Experimental): PMN310 1400 mg or placebo administered as a 60-minute infusion.
  Interventions: Drug: PMN310; Drug: Placebo

INTERVENTIONS:
Drug: PMN310 — A humanized immunoglobulin G1 (IgG1) monoclonal antibody
Drug: Placebo — 0.9% NaCl 100 mL

SUMMARY:
This Phase 1b study aims to evaluate the safety, tolerability, pharmacokinetics, pharmacodynamics, and preliminary efficacy of multiple IV infusions of PMN310 in patients with early Alzheimer's disease.

DETAILED DESCRIPTION:
This study is a Phase 1b, randomized, double-blind, placebo controlled, multi-ascending dose study of repeat doses of PMN310 to evaluate the safety, tolerability, PK, PD, and preliminary efficacy of multiple intravenous infusions of PMN310 in patients with early Alzheimer's disease. This study will evaluate 3 dose levels (350 mg, 700 mg, and 1400 mg are planned). Patients will be randomly assigned 3:1, PMN310: placebo.

Each patient will receive PMN310 or placebo once every 28 days for a total of 12 infusions.

ELIGIBILITY:
Inclusion Criteria:

1. Patient and caregiver provide written informed consent.
2. Ambulatory male or female ≥ 50 years of age with adequate visual and auditory abilities to perform the cognitive and functional assessments in the opinion of the Investigator.
3. Meets all of the following clinical criteria for mild cognitive impairment (MCI) due to AD or mild AD dementia at Screening:

   1. National Institute on Aging-Alzheimer's Association criteria for MCI due to AD or mild AD dementia (Stage 3 and 4)
   2. Global Clinical Dementia Rating (CDR) of 0.5 1.0 and memory box score ≥ 0.5 at Screening and Baseline
   3. Objective impairment in episodic memory as indicated by at least 1 standard deviation (SD) below age-adjusted mean in the Wechsler Memory Scale IV-Logical Memory (subscale) II
   4. MMSE score between ≥ 20 and 28 inclusive at Screening, and
   5. Either a positive amyloid PET scan within 6 months of Screening consistent with AD, or a positive amyloid PET during Screening.
4. Body mass index between 18.5 and 35 kg/m2 inclusive.
5. Patients of childbearing potential must meet the following criteria:

   1. Male and female patients with reproductive potential must be willing to use an approved double barrier contraceptive method (e.g., condom plus intrauterine device, condom plus hormonal contraception, or double barrier device) during and for 120 days after the last dose of study drug
   2. Females of childbearing potential must have a negative serum pregnancy test during Screening, a negative urine pregnancy test prior to each dose, and not currently be breastfeeding.
6. Patients of non-childbearing potential must meet 1 of the following:

   1. Post-menopausal female (i.e., 12 consecutive months of spontaneous amenorrhea, age > 51 years, and follicle-stimulating hormone > 30 mIU/mL)
   2. Surgically sterile (i.e., bilateral oophorectomy or hysterectomy).
7. Has a reliable caregiver who agrees to accompany the patient at study visits, accurately report patient's status, provide feedback on functional and safety assessments, and ensure compliance to study requirements.
8. Confirmed to have acceptable venous access for blood collections and IV administration of study drug (i.e., PMN310 or placebo).
9. Patients taking Food and Drug Administration-approved acetylcholinesterase inhibitors or memantine are allowed as long as the dose has been stable for at least 3 months prior to Screening.

Exclusion Criteria:

1. Living in a continuous care or long-term care nursing facility. Patients in outpatient living at home or in an assisted living facility are eligible for the study.
2. Medical or neurological condition (other than AD; i.e., Parkinson's disease, Huntington's disease, frontal temporal dementia, dementia with Lewy bodies) judged to be contributing to the patient's cognitive impairment.
3. Laboratory and electrocardiogram (ECG) abnormalities:

   1. QT (QTcF) interval > 450 msec (males) or > 470 msec (females) during Screening
   2. Alanine aminotransferase ≥ 2 × upper limit of normal (ULN); aspartate aminotransferase ≥ 2 × ULN; total bilirubin ≥1.5 × ULN during Screening
   3. Creatinine clearance < 30mL/min during Screening.
4. In the opinion of the Investigator, any clinically significant current or relevant history of physical or psychiatric illness (including suicidal risk, ideation, behavior, or suicide attempts), any medical disorder that may require treatment or make the patient unlikely to fully complete the study, or any condition that presents undue risk from the investigational product or procedures.
5. Clinically significant recurrent disease or unstable disease that could affect the action, absorption, or disposition of the investigational product, or could affect clinical or laboratory assessments, such as (but not limited to) the following:

   1. History of unstable angina, myocardial infarction, chronic heart failure, or clinically significant conduction abnormalities within 1 year prior to Screening
   2. Indication of clinically significant impairment of renal or liver function, including hepatitis B surface antigen, or hepatitis C virus antibody at Screening
   3. Poorly managed hypertension (systolic > 160 mmHg and/or diastolic > 95 mmHg) or hypotension (systolic < 90 mmHg and/or diastolic < 60 mmHg). Two repeated assessments during Screening are allowed
   4. Known uncontrolled diabetes defined by hemoglobin A1c > 7.5 or insulin dependent diabetes.
6. Experienced a significant systemic illness, as judged by the Investigator, within 30 days of the first dose of study drug.
7. Seizure in the 3 years prior to Screening.
8. History of a clinically significant medical condition that would interfere with the patient's ability to comply with study instructions, would place the patient at increased risk, or might confound the interpretation of the study results.
9. History of prior malignancy (except adequately treated non-melanoma skin cancer or carcinoma in situ of the cervix).
10. Brain MRI with evidence of any of the following findings at Screening: >4 microhemorrhages; > 1 lobar microhemorrhage, area of superficial siderosis; subarachnoid hemorrhage; any other hemorrhage > 10 mm; > 2 lacunar infarcts or cortical infarct; subjects with severe perivascular spaces or with white matter hyperintensities in a multisport pattern will require PI review prior to inclusion.
11. History of stroke or transient ischemic attack within 12 months prior to Screening.
12. Contraindication to PET or brain MRI.
13. Negative PET scan with any amyloid-targeting ligand within 6 months of Screening or during Screening.
14. Pregnant or breastfeeding.
15. History of alcohol abuse and/or other substance abuse within 12 months prior to dosing with study drug.
16. Positive test for alcohol (using an alcohol breath test) or illicit drugs of abuse at Screening.
17. Documented history of human immunodeficiency virus antibody.
18. Coronavirus disease 2019 (COVID-19) infection within 2 weeks of Screening or ongoing symptoms of COVID-19 at Screening.
19. Currently receiving an anti-amyloid treatment, either marketed (aducanumab, lecanemab, donanemab) or investigational or has received anti amyloid therapy within 9 months prior to Screening. In the case of investigational treatment, those known to have received placebo will not be excluded.
20. Contraindication to undergoing lumbar puncture (LP) including: sensitivity to local anesthetic, international normalized ratio (INR) > 1.4 or other coagulopathy, platelet cell count of < 120,000/µL, infection at the desired LP site, current use of anti-coagulant medication except for low dose aspirin, degenerative arthritis, spinal scoliosis, back surgery, suspected increased intracranial pressure on history or neurologic exam, non-communicating hydrocephalus or intracranial mass, or prior history of spinal mass or trauma and/or other known clinically significant spinal abnormalities.
21. Donated blood or blood products (e.g., plasma, platelets) within 56 days prior to first dose of study drug.
22. Received an investigational active agent (e.g., not placebo) within the last 30 days or 5 half-lives, whichever is longer (if known).
23. Known history of severe allergic reaction or hypersensitivity to any components of the PMN310 infusion.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 144 (Estimated)
Dates: Start 2024-12-13 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Safety and tolerability of PMN310 following repeat intravenous infusions of PMN310 | Up to Day 365
  Number and severity of adverse events
Biomarker response to PMN310 following repeat intravenous infusions of PMN310 | Up to Day 365
  Mean change in plasma p-tau217 in response to repeat intravenous infusions of PMN310
Safety and tolerability of PMN310 following repeat intravenous infusions of PMN310 | Up to Day 365
  Percent of patients with symptomatic and/or non symptomatic amyloid-related imaging abnormalities
Biomarker response to PMN310 following repeat intravenous infusions of PMN310 | Up to Day 365
  Mean change in amyloid PET in response to repeat intravenous infusions of PMN310

SECONDARY OUTCOMES:
Pk profile of PMN310 with repeat dosing | Up to Day 365
  Serum PK parameter area under the curve to the end of the dosing period (AUCtau)
Assessment of the immunogenicity of PMN310 following repeat intravenous infusions | Up to Day 365
  Immunogenicity of PMN310 - anti-drug antibodies (ADAs) in serum
Assessment of biomarker response to PMN310 | Up to Day 365
  Mean change from baseline for ABeta PET
Assessment of cortical and hippocampal volume | Up to Day 365
  Mean change from Baseline in cortical and hippocampal volume
Preliminary efficacy of repeat doses of PMN310 on CDR-SB | Up to Day 365
  Mean change from Baseline in Clinical Dementia Rating Scale-Sum of Boxes (CDR-SB)
Pk profile of PMN310 with repeat dosing | Up to Day 365
  Serum PK parameter concentration 4 weeks post-dose (C4W)
Pk profile of PMN310 with repeat dosing | Up to Day 365
  Serum PK parameter maximum observed concentration (Cmax)
Pk profile of PMN310 with repeat dosing | Up to Day 365
  Serum PK parameter trough concentration (Ctrough)
Pk profile of PMN310 with repeat dosing | Up to Day 365
  Serum PK parameter time to reach maximum observed concentration (Tmax)
Pk profile of PMN310 with repeat dosing | Up to Day 365
  Concentration of PMN310 in CSF at selected timepoints
Assessment of biomarker response to PMN310 | Up to Day 365
  Mean change from baseline for imaging
Assessment of biomarker response to PMN310 | Up to Day 365
  Mean change from baseline for plasma biomarkers
Assessment of biomarker response to PMN310 | Up to Day 365
  Mean change from baseline for CSF biomarkers
Preliminary efficacy of repeat doses of PMN310 on ADAS-Cog 14 | Up to Day 365
  Mean change from Baseline in Alzheimer's Disease Assessment Scale-Cognition 14 item (ADAS-Cog 14)
Preliminary efficacy of repeat doses of PMN310 on ADCS-ADL | Up to Day 365
  Mean change from Baseline in Alzheimer's Disease Cooperative Study-Activities of Daily Living (ADCS-ADL)
Preliminary efficacy of repeat doses of PMN310 on iADRS | Up to Day 365
  Mean change from Baseline in Integrated Alzheimer's Disease Rating Score (iADRS)
Preliminary efficacy of repeat doses of PMN310 on CGI Scale | Up to Day 365
  Mean change from Baseline in Clinical Global Impressions (CGI) Scale
Preliminary efficacy of repeat doses of PMN310 on MMSE | Up to Day 365
  Mean change from Baseline in Mini-Mental State Examination (MMSE)

CONTACTS AND LOCATIONS:
Locations (22):
- United States (22):
  - Irvine Center for Clinical Research, Irvine, California
  - Healthy Brain Research, Long Beach, California
  - JEM Research Institute, Atlantis, Florida
  - Quantum Laboratories, Deerfield Beach, Florida
  - Brain Matters Research, Delray Beach, Florida
  - Finlay Medical Research, Miami, Florida
  - Gonzalez MD and Aswad MD Health Services, Optimus U Corp, Miami, Florida
  - Renstar Medical Research, Ocala, Florida
  - Charter Research, Orlando, Florida
  - Alzheimer's Research and Treatment Center, Stuart, Florida
  - Charter Research, The Villages, Florida
  - Alzheimer's Research and Treatment Center, Wellington, Florida
  - Conquest Research, LLC, Winter Park, Florida
  - Columbus Memory Center, LLC, Columbus, Georgia
  - CenExel iResearch, LLC, Decatur, Georgia
  - Headlands Eastern MA LLC, Plymouth, Massachusetts
  - Advanced Memory Research Institute of NJ, Toms River, New Jersey
  - Alzheimer's Disease Research Center, Albany, New York
  - Flourish Research, Matthews, North Carolina
  - Neuro Behavioral Clinical Research, Inc., North Canton, Ohio
  - Keystone Clinical Studies, LLC, Plymouth Meeting, Pennsylvania
  - Kerwin Medical Center, Dallas, Texas